CLINICAL TRIAL: NCT03654079
Title: Patient Centered Simulation For Labor and Delivery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB00052749
Record Dates: First submitted 2018-08-28; First posted 2018-08-31 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy Related
Keywords: Simulation; Pregnancy; Labor and Delivery; Childbirth

STUDY DESIGN:
Intervention Model Description: Women in Centering Pregnancy groups at Wake Forest School of Medicine's Obstetrics (OB) and Gynecology (GYN) department will be recruited and sequentially assigned to participate in simulations or serve as controls.
Who Masked: Outcomes Assessor
Masking Description: Group assignment will be removed from the data set prior to analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation Arm (Active Comparator): Subjects in this arm will participate in Interventions (In- Utero Simulation, Cesarean Section Simulation, and Pushing Simulation).
  Interventions: Other: Simulation
- Control Arm (No Intervention): Subjects in this arm will not participate in any simulations.

INTERVENTIONS:
Other: Simulation — Participants assigned to the intervention group will participate in the following simulations: 1) the process that may occur if a baby has a significant drop in heart rate during labor, 2) the process of moving from the labor bed to the transport stretcher and on to the operating room in the event that a woman needs a cesarean delivery, 3) the pushing process after a woman becomes completely dilated
  Arms: Simulation Arm

SUMMARY:
Patient satisfaction is an important outcome in the evaluation and development of healthcare services. Studies have identified tools that successfully measure women's childbirth experiences, and have shown that multidimensional measures of women's satisfaction in labor and delivery provides a richer and diverse perspective on women's experiences of intrapartum care. Childbirth experience can have significant effects, both positive and negative, on women's immediate and long term health outcomes. Patients with negative experiences surrounding childbirth have been shown to have significant fear surrounding the labor and delivery experience that negatively impact subsequent deliveries. Often fear is worsened by a lack of knowledge of what to expect during labor. Women enrolled in this study will simulate some of the potentially stressful experiences that commonly occur during labor to determine if doing so decreases a woman's fear and anxiety about labor and delivery.

DETAILED DESCRIPTION:
Patient satisfaction is an important outcome in the evaluation and development of healthcare services. Studies have identified tools that successfully measure women's childbirth experiences, and have shown that multidimensional measures of women's satisfaction in labor and delivery provides a richer and diverse perspective on women's experiences of intrapartum care. Childbirth experience can have significant effects, both positive and negative, on women's immediate and long term health outcomes. Patients with negative experiences surrounding childbirth have been shown to have significant fear surrounding the labor and delivery experience that negatively impact subsequent deliveries. Often fear is worsened by a lack of knowledge of what to expect during labor. Women enrolled in this study will simulate some of the potentially stressful experiences that commonly occur during labor to determine if doing so decreases a woman's fear and anxiety about labor and delivery. Women in Centering Pregnancy groups will be approached and assigned to either the intervention or control arm by Centering Pregnancy group. Those in the intervention arm will participate in simulations in the following areas: 1) In-Utero Resuscitation Simulation: the process that may occur if a baby has a significant drop in heart rate during labor, 2) Cesarean Section Simulation: the process of moving from the labor bed to the transport stretcher and on to the operating room in the event that a laboring woman needs a cesarean delivery, 3) Pushing Simulation: the pushing process after a laboring woman becomes completely dilated. Those in the control arm will not receive this education. All patient will complete a modified Childbirth Experience Questionnaire the day after delivery. Responses will be compared between the woman that participated in the simulations to women who did not participate in simulations.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous pregnant women
* In third trimester

Exclusion Criteria:

• Not planning on delivering with Wake Forest School of Medicine OB/GYN

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregnant women are eligible for this study
Enrollment: 50 (Estimated)
Dates: Start 2026-07 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Childbirth Experience Questionnaire (CEQ) | After delivery, up to 2 weeks
  Childbirth Experience Satisfaction will be measured by the CEQ a 24 item questionnaire. For 19 of the items the response format is a 4-point Likert Scale and three of the items are assessed using a visual analogue scale (VAS). The VAS-scales scores were transformed to categorical values, 0-40 = 1, 41-60 = 2, 61-80 = 3 and 81-100 = 4. Total score 24-92. Higher scores indicate better childbirth experience

CONTACTS AND LOCATIONS:
Overall Officials: Joshua F Nitsche, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest Baptist Health Downtown Health Plaza, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rudman A, El-Khouri B, Waldenstrom U. Women's satisfaction with intrapartum care - a pattern approach. J Adv Nurs. 2007 Sep;59(5):474-87. doi: 10.1111/j.1365-2648.2007.04323.x. Epub 2007 Jul 20. PMID 17645495
- [Background] Nilver H, Begley C, Berg M. Measuring women's childbirth experiences: a systematic review for identification and analysis of validated instruments. BMC Pregnancy Childbirth. 2017 Jun 29;17(1):203. doi: 10.1186/s12884-017-1356-y. PMID 28662645
- [Background] Nilsson C, Lundgren I, Karlstrom A, Hildingsson I. Self reported fear of childbirth and its association with women's birth experience and mode of delivery: a longitudinal population-based study. Women Birth. 2012 Sep;25(3):114-21. doi: 10.1016/j.wombi.2011.06.001. Epub 2011 Jul 20. PMID 21764400
- [Background] World Health Organization . WHO Statment: The prevention and elimiation of disrespect and abuse during facility-based childbirth. 2014.
- [Background] Finnbogason, Christine. "Experiences and Satisfaction with Intrapartum Care: A Comparison of Normal Weight Women and Obese Women." University of Manitoba, University of Manitoba, 2016, pp. 149-154.